CLINICAL TRIAL: NCT04070352
Title: Evaluation of Fidaxomicin in the Treatment of Clostridium Difficile Infection (CDI)
Status: Withdrawn | Type: Observational
Why Stopped: no patients enrolled
Sponsor: University of Pittsburgh (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO18110022
Record Dates: First submitted 2019-08-13; First posted 2019-08-28 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2022-06

CONDITIONS: Clostridium Difficile Infection (CDI)
MeSH Terms: conditions — Clostridium Infections | interventions — Fidaxomicin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All discarded biological samples collected as part of the patient's clinical care to include blood, urine, BAL, tissue, etc. Additionally a blood sample is obtained for genetic testing and CDI analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- clostridium difficile infection (CDI): This is a pilot project. Data from electronic medical records will be collected on all patients diagnosed with clostridium difficile infection and who are receiving fidaxomicin as part of their treatment. A total of 50 patients will be enrolled
  Interventions: Drug: Fidaxomicin

INTERVENTIONS:
Drug: Fidaxomicin — patients who are receiving fidaxomicin are enrolled into the study, blood is obtained for analysis, EMR and outcome data collected regarding their CDI
  Other Names: clostridium difficile infection

SUMMARY:
This is a single center collection of discarded biological samples and electronic medical review (EMR) data on patients who are hospitalized with clostridium difficile infections and treated with Fidaxomicin

DETAILED DESCRIPTION:
This single site study will be a clinical research data base of patients hospitalized and diagnosed with Clostridium difficile infection (CDI), treated with Fidaxomicin and willing to allow us to collect discard biological samples for testing and analysis in the investigators lab. An additional blood sample will be obtained if a clinically indicated bronchoscopy is performed as to measure the amount of medication in the BAL. We will also complete a medical record review will also occur.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age
2. Currently an inpatient at UPMC Presbyterian
3. Diagnosed with an CDI
4. Being treated with Fidaxomicin

Exclusion Criteria:

not meeting entry criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with CDI and treated with fidaxomicin and seen at PUH
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
risks factors | "1 year"
  Incidence of death as indicated in medical record

SECONDARY OUTCOMES:
CDI episodes | "1 year"
  quantified by number of stools in a day as reported in medical record

CONTACTS AND LOCATIONS:
Overall Officials: Cornelius Clancy, MD, Principal Investigator — UPMC and PITT
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
This is a pilot project. research data/samples may be shared with investigators conducting other research; this information will be shared without identifiable information. If such will occur appropriate regulatory documentation such as DUA or MTA's will be put in place prior to sharing of data and biological samples

REFERENCES:
- [Result] Pant C, Anderson MP, O'Connor JA, Marshall CM, Deshpande A, Sferra TJ. Association of Clostridium difficile infection with outcomes of hospitalized solid organ transplant recipients: results from the 2009 Nationwide Inpatient Sample database. Transpl Infect Dis. 2012 Oct;14(5):540-7. doi: 10.1111/j.1399-3062.2012.00761.x. Epub 2012 Jun 22. PMID 22726461
- [Result] Heimann SM, Cruz Aguilar MR, Mellinghof S, Vehreschild MJGT. Economic burden and cost-effective management of Clostridium difficile infections. Med Mal Infect. 2018 Feb;48(1):23-29. doi: 10.1016/j.medmal.2017.10.010. Epub 2018 Jan 12. PMID 29336929
- [Result] Nathwani D, Cornely OA, Van Engen AK, Odufowora-Sita O, Retsa P, Odeyemi IA. Cost-effectiveness analysis of fidaxomicin versus vancomycin in Clostridium difficile infection. J Antimicrob Chemother. 2014 Nov;69(11):2901-12. doi: 10.1093/jac/dku257. Epub 2014 Aug 5. PMID 25096079
- [Result] Nguyen CT, Li J, Anders S, Garcia-Diaz J, Staffeld-Coit C, Hand J. Comparison of outcomes with vancomycin or metronidazole for mild-to-moderate Clostridium difficile associated diarrhea among solid organ transplant recipients: A retrospective cohort study. Transpl Infect Dis. 2018 Jun;20(3):e12867. doi: 10.1111/tid.12867. Epub 2018 Mar 30. PMID 29512244
- [Result] Cornely OA, Watt M, McCrea C, Goldenberg SD, De Nigris E. Extended-pulsed fidaxomicin versus vancomycin for Clostridium difficile infection in patients aged >/=60 years (EXTEND): analysis of cost-effectiveness. J Antimicrob Chemother. 2018 Sep 1;73(9):2529-2539. doi: 10.1093/jac/dky184. PMID 29800295